CLINICAL TRIAL: NCT06232083
Title: A Multi Tumor, Open Phase I Clinical Study on the Progression of First-line Anti-tumor Therapy Using Cardonizumab Combined With Pulsed Low-dose Rate External Irradiation (PLDR)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhou peijie-2024ky-05
Record Dates: First submitted 2024-01-16; First posted 2024-01-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer; Esophageal Cancer; Cervical Cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLDR+Cadonilimab (Experimental): 1. PLDR: 40Gy/20f; GTV is the recurrence or metastasis lesion with clear imaging (the radiotherapy lesion is determined by the researcher, and the first-line treatment is preferred for the advanced lesion). CTV is the appropriate expansion of GTV by 0.5cm-0.7cm, including the related lymphatic drainage area (such as neck and pelvic cavity) if necessary.
  2. ICB was performed during the external irradiation of PLDR, and cadunizumab 6mg/kg was given for 2 weeks; After the external irradiation of PLDR, cardunilimab was maintained at the dose of 10mg/kg for 3 weeks. Maintenance treatment for 2 years.
  Interventions: Radiation: PLDR+Cardunizumab

INTERVENTIONS:
Radiation: PLDR+Cardunizumab — Application of PLDR external irradiation combined with Cardunizumab in recurrent lung cancer, esophageal cancer and cervical cancer.

SUMMARY:
At present, the treatment methods for recurrent cancers are very limited. The immune checkpoint inhibitors (ICBs) is a promising new directions for recurrent lung cancer/ esophageal cancer / cervical cancer, but the clinical response rate is insufficient. Pulse low-dose rate radiotherapy (PLDR) is a new technology in recent years, which uses continuous pulse low-dose rate irradiation to induce hypersensitivity in tumors, and its clinical safety has been verified. Compared to conventional radiotherapy, PLDR has advantages in protecting the lymphatic system and relieving the immune barrier, but it is still unclear whether it can improve the efficacy of ICB. This project aims to combine PLDR with ICB to explore new strategies for recurrent patients.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all the following criteria to be enrolled:

1. The subjects voluntarily joined the study, signed informed consent, had good compliance and were willing to cooperate with the follow-up;
2. There is no limit for men and women, ranging in age from 18 to 75 years old (including 18 and 75 years old);
3. Pathologically confirmed esophageal cancer, lung cancer or cervical cancer;
4. The expected survival time was more than 3 months;
5. Recurrent or metastatic patients with previous treatment progress;
6. ECoG 0-2 points;
7. According to RECIST 1.1 standard, there was at least one extracranial measurable lesion;
8. The laboratory test results within one week before enrollment meet the following conditions: 1) blood routine: HGB≥90g/L； WBC ≥ 4.0 × 109/L; Neut ≥ 2.0 × 109/l; PLT ≥ 100 × 109/l; 2) Blood biochemistry: TBIL ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN (ALT and AST ≤ 5 × ULN in patients with liver metastasis); Bun and Cr ≤ 1.5 × ULN and creatinine clearance rate ≥ 50 ml/min; 3) The results of echocardiography within two weeks before admission were consistent: left ventricular ejection fraction (LVEF)>50%;
9. The coagulation function was normal without active bleeding and thrombosis;
10. Patients without contraindications to radiotherapy;
11. The pregnancy test of patients of childbearing age was negative, and they voluntarily took effective and reliable contraceptive measures during the test;
12. Subjects who have received anti-tumor treatment in the past should not be enrolled until the toxicity of previous treatment has stabilized and returned to the baseline level (except for the residual hair loss effect) or the CTCAE V5.0 score ≤ 1.

Exclusion criteria

If the patient meets any of the following conditions, he cannot be selected:

1. Patients with malignant tumors other than esophageal cancer, lung cancer and cervical cancer;
2. Patients with other active malignant tumors in the first 5 years of randomization, such as squamous cell carcinoma of the skin, basal cell carcinoma of the skin, superficial bladder cancer, and breast cancer in situ, except those with locally curable tumors that have been cured;
3. Patients who had participated in clinical trials of other drugs within 4 weeks before enrollment, and who had received radiotherapy for the target area within 4 weeks before entering this study, were vaccinated with live attenuated vaccine within 4 weeks before the first administration or during the study period;
4. Arteriovenous thrombosis events occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, etc;
5. Receiving any other anti-tumor treatment at the same time;
6. Those who are known to have a history of allergy to the drug components of this protocol have a history of telangiectatic ataxia or other radiation hypersensitivity;
7. Subjects with active infectious diseases;
8. Subjects with any severe and/or uncontrolled disease;
9. Female patients during pregnancy and lactation, female patients with fertility and positive baseline pregnancy test;
10. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study (including but not limited to severe hypertension, severe pulmonary dysfunction/disease and severe diabetes that cannot be controlled by drugs);
11. Having a clear history of neurological or mental disorders, including epilepsy or dementia, and unable to cooperate with the radiotherapy process;
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
13. Diagnosed with immune deficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy, and suffering from active or recurrent autoimmune diseases, except for vitiligo, alopecia, psoriasis or eczema that do not require systematic treatment; Hypothyroidism caused by autoimmune thyroiditis only needs a stable dose of hormone replacement therapy; Type I diabetes requiring only a stable dose of insulin replacement therapy;
14. Have active or documented inflammatory bowel disease (such as Crohn's disease, ulcerative colitis), and active diverticulitis. The clinical manifestations of gastrointestinal obstruction, or the need for conventional parenteral fluid infusion, parenteral nutrition or indwelling gastric tube;
15. There were symptomatic central nervous system (CNS) metastasis, leptomeningeal metastasis or spinal cord compression caused by metastasis before signing the informed consent. Those without clinical symptoms, who have clinical and/or imaging evidence indicating stable condition, and who stop corticosteroids and anticonvulsant drugs for at least 2 weeks can participate in the study;
16. At present, there are patients with effusion in the third space who need repeated puncture and drainage and other local treatment with poor clinical control;
17. Subjects with any of the following cardiovascular diseases were excluded:

    1. Myocardial infarction, unstable angina pectoris, pulmonary embolism, acute/persistent myocardial ischemia, cerebrovascular accident, transient ischemic attack, or other arteriovenous thrombosis, embolism or ischemic events with clinical significance/requiring drug treatment intervention occurred within 6 months before the first administration;
    2. Previous and/or current NYHA III-IV congestive heart failure;
    3. Previous and/or current severe arrhythmias requiring medical treatment;
    4. Before the first administration, 12 lead ECG showed that the mean QT interval (QTCF)>470 Ms.
18. The investigator believes that the patient is not suitable for any other circumstances in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 month post PLDR external irradiation
  Objective response rate，The proportion of patients whose tumor volume shrinks by 30% and can be maintained for more than four weeks, which is the sum of complete remission and partial remission (CR+PR)

SECONDARY OUTCOMES:
TEAE | 6 month post PLDR external irradiation
  Treatment Emergent Adverse Event

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, British Columbia, China

IPD SHARING:
Plan to Share IPD: Undecided